CLINICAL TRIAL: NCT02616978
Title: Retrospective Study on the Use of CEFALY® Device During Migraine Attacks
Status: Completed | Type: Observational
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: 50214
Record Dates: First submitted 2015-11-19; First posted 2015-11-30 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an Internet survey to collect data on the use of the Cefaly device to treat migraine attacks in regular Cefaly users.

DETAILED DESCRIPTION:
About 1000 CEFALY users, having the device since more than one year and having reordered electrodes in the last year, will be invited to participate to an Internet survey. This survey contains at most 8 questions, and data will be collected completely anonymously. Questions concern the use or not of the CEFALY during migraine attacks, the number of treated attacks and the number and type of acute anti-migraine drugs that were avoided thanks to the use of the CEFALY.

ELIGIBILITY:
Inclusion Criteria:

* Subjects using Cefaly device regularly for more than a year identify by reordering of electrodes during the last year.
* History of likely episodic or chronic migraine with or without aura diagnosed by a physician

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French speaking patients in Belgium, Switzerland and France, having ordered new electrodes during the last year will be identified as regular users.
Sampling Method: Non-Probability Sample
Enrollment: 807 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Monthly number of acute drug intake avoided when using Cefaly to treat a migraine attack | Maximum 1 year
  On average, mean number of anti-migraine acute drug intake avoided per month per patient in regular Cefaly users, based on self reported average monthly number of attacks and percentage of attacks treated successfully with the Cefaly

SECONDARY OUTCOMES:
Proportion of Cefaly users that report using also the device to treat migraine attacks | Maximum 1 year
  Percentage of regular Cefaly users using the device to treat attacks
Proportion of migraine attacks treated with the Cefaly device | Maximum 1 year
  Percentage of migraine attacks treated with the Cefaly device by the Cefaly users
Proportion of migraine attacks for which the use of the Cefaly device generate a reduction of drug intake | Maximum 1 year
  Percentage of migraine attacks treated with the Cefaly device and for which the acute anti-migraine drug intake is reduced thanks to the Cefaly

REFERENCES:
- [Result] Penning S, Schoenen J. A survey on migraine attack treatment with the CEFALY(R) device in regular users. Acta Neurol Belg. 2017 Jun;117(2):547-549. doi: 10.1007/s13760-017-0757-z. Epub 2017 Feb 9. No abstract available. PMID 28185179